CLINICAL TRIAL: NCT06112626
Title: Chlorhexidine Gluconate Bathing Education Video Intervention Among Hospitalized Patients: A Pragmatic Cluster Randomized Clinical Trial
Brief Title: Chlorhexidine Gluconate Bathing Education Video Among Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Massachusetts General Hospital (Other); Indiana University Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00112033
Record Dates: First submitted 2023-10-10; First posted 2023-11-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group: In addition to the current educational document available for CHG bathing, patients in the intervention group would be provided access to a CHG bathing video through multiple avenues (QR codes placed in the room/unit, video provided on unit iPads). Nurses will be instructed to provide QR codes to patients to scan and watch the video. Patients can scan the QR code using their own smart device or through unit-based iPads. After viewing the video, there is another QR code to scan that goes to a short patient survey.
  Interventions: Behavioral: CHG Skin Treatment Video
- Control Group (No Intervention): Control Group: Patients in the control group would have access to the current education available (patient education document) - usual care

INTERVENTIONS:
Behavioral: CHG Skin Treatment Video — Short CHG skin treatment video that reviews the rationale/importance of CHG bathing, and the appropriate process for bathing
  Arms: Intervention Group

SUMMARY:
Chlorhexidine gluconate (CHG) bathing is an effective intervention to reduce hospitalized patient's risk of acquiring a central line-associated bloodstream infection (CLABSI). While daily CHG bathing for hospitalized patients is widely supported in the literature, patient adherence with this practice is suboptimal. Written and verbal information is provided to patients by nursing staff regarding the importance of CHG bathing and the correct usage of the CHG cloths; however, these methods can be hindered by literacy and language barriers. Medical videos have become popular avenues to provide necessary education to patients, and have been shown to improve patient-reported outcomes. Whereas the benefits of educational videos has been described in previous studies on advanced care planning and postoperative quality of life, they have not been described for CHG bathing. In this study, we aim to provide education (including the rationale/importance of CHG bathing, and the appropriate process for bathing) through the use of a short video provided to hospitalized patients. The purpose of this study is to evaluate the use of medical videos to educate patients on CHG bathing while hospitalized in the inpatient setting.

DETAILED DESCRIPTION:
For this study, approximately 16 inpatient units will be included; 8 will be randomized to the intervention (access to patient-facing CHG video) with the remaining units continuing with usual care (providing education via verbal/written information). All patients who require a CHG bath would be eligible to participate.

Intervention Group: In addition to the current educational document available for CHG bathing, patients admitted to the intervention units will be provided access to a CHG bathing video through multiple avenues (QR codes placed in the room/unit, video provided on unit iPads). Nurses will be instructed to provide QR codes to patients to scan and watch the video. Patients can scan the QR code using their own smart device or through unit-based iPads. After viewing the video, patients will be directed to scan a separate QR code to complete a voluntary questionnaire.

Control Group: Patients in the control group would have access to the current education available (patient education document) - usual care

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an intervention unit who require a CHG skin treatment

Exclusion Criteria:

* CHG allergy
* Patients on comfort care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a documented chlorhexidine gluconate bath documentation compliance | Up to 12 months
  Compliance with documenting CHG bath treatment in the electronic health record; measured via a report from the electronic health record

SECONDARY OUTCOMES:
Rate of central line associated bloodstream infections per 1000 central line days | Up to 12 months
  Central line associated bloodstream infection rate per 1000 patient days, measured by standard National Healthcare Safety Network (NHSN) criteria by the hospital's infection prevention departments
Patient use of CHG skin treatment video | 4 weeks
  number of patients who opened the video, percentage of patients who opened the video (# of video views / total # of patients admitted to the unit per month), percentage of the video viewed
Patient-centered outcome questionnaire | 4 weeks
  Patients' perceptions of: how helpful they found the video; if they are likely to participate in CHG skin treatments; how comfortable they were watching the video

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Hospital, Durham, North Carolina
  - WakeMed Health and Hospitals, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No